CLINICAL TRIAL: NCT01048827
Title: A Phase I Study of Targeted, Dose-Escalated Intravenous Busulfan and Bolus Etoposide as Preparative Therapy for Patients With Acute Myeloid Leukemia Undergoing Autologous Stem Cell Transplantation
Brief Title: Targeted, Dose-Escalation Busulfan-Etoposide as Prep Regimen
Acronym: Busulfan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 82516; NCT00824525 (obsolete NCT alias)
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; autologous transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- experimental (Experimental): dose-escalation Busulfan
  Interventions: Drug: Busulfan

INTERVENTIONS:
Drug: Busulfan — 1. 1250 uMol*min (AUC to time 6 hrs)^
  2. 1400 uMol*min (AUC to time 6 hrs
  3. 1550 uMol*min (AUC to time 6 hrs)^

SUMMARY:
Busulfan and etoposide have been used as preparative therapy for autoSCT (stem cell transplant) in adults with acute myeloid leukemia (AML) at UCSF for the past 10 years. Over this period and together with collaborative transplant centers, over 200 patients have received this treatment. By intent-to-treat analysis, and with median follow-up of 7.0 years, the 5-year DFS is 55%. The current protocol will utilize the combination of IV Busulfan (BU) and etoposide. The busulfan dose will be escalated amongst 3 targeted dose levels. All targeted dose levels represent higher busulfan dosing than standard myeloablative dosing, with the lowest dose being approximately 14% higher than standard. Busulfan levels will be monitored after the first, fourth and twelfth doses. Dose adjustments will be made "in real time" based on AUC levels determined from the first and fourth doses. This strategy of busulfan monitoring and dose adjustment has improved the therapeutic widow of BU in previous clinical trials.

The current protocol will utilize the combination of intravenous busulfan and etoposide. The busulfan dose will be escalated amongst 3 targeted dose levels (area under the curve (AUC) levels at time 6 hours of 1250 uMol*min, 1400 uMol*min and 1550 uMol*min). All targeted dose levels represent higher busulfan dosing than standard myeloablative dosing with the lowest dose (1250 uMol*min) being approximately 14% higher than standard. In the absence of dose-limiting toxicity, cohorts of 4-6 patients will be treated at each dose level and 10 additional patients will be treated at the maximum tolerated dose (MTD) to confirm safety. The busulfan dosing will begin at 1 mg/kg based on historical plasma levels obtained from patients receiving BU at a starting dose of 0.8 mg/kg at UCSF Medical Center.

The highest dose level proposed for this study will exceed the reported toxic level for busulfan in the alloSCT setting. Patients will be followed closely for toxicity and strict stopping rules have been included. Eligibility criteria will exclude patients with prior history of hepatotoxicity or viral hepatitis. Potential hepatotoxic agents will not be allowed just prior to and during the busulfan dosing period. In addition, patients who experience hepatotoxicty during pre-transplant mobilization therapy may be excluded from receiving dose-escalated busulfan therapy. Every attempt will be made to prevent or avoid hepatotoxicity.

DETAILED DESCRIPTION:
TREATMENT: STEP 1 - CONSOLIDATION CHEMOTHERAPY

* Etoposide 10 mg/kg IV continuous infusion over 24 hrs for 4 days (total course dose 40 mg/kg). Dose should be based on corrected weight, calculated as follows: Ideal + 25% of the difference between actual and ideal weight. If actual is less than ideal weight use actual weight. Etoposide infusion should be mixed in normal saline at a concentration of 0.4-0.5 mg/ml. The infusion volume will be approximately 1.39 ml/kg/hour and should be rounded to the nearest 500-1000 ml and infused through a central venous catheter.
* Cytarabine (ara-C) 2,000 mg/m2 IV over 2 h q 12 h x 8 doses Days 1-4. Cytarabine dosage should be based on corrected weight, calculated as follows: Ideal weight + 25% of the difference between actual and ideal weight. If actual weight is less than ideal weight, use actual weight.Begin concurrent with etoposide infusion. Cytarabine doses should be mixed in 250 ml of D5W.

To prevent neurotoxicity from high-dose cytarabine (HDAC), cytarabine doses will be adjusted according to renal function. The dose of cytarabine will be reduced to 1000 mg/m2/dose if creatinine is 1.5-1.9 mg/dL or if there is an increase from baseline creatinine at start of cytarabine of 0.6-1.1 mg/dL (example: baseline creatinine 0.8 mg/dL increase to 1.4 mg/dL (difference of 0.6 mg/dL)), decrease cytarabine to 1000 mg/m2/dose.The dose of cytarabine will be reduced to 100 mg/m2/dose if creatinine > 2.0 mg/dL or if there is an increase from baseline > 1.2 mg/dL.Cytarabine will be discontinued immediately for any clinical evidence of cerebellar neurotoxicity (dysarthria, dysmetria, gait disturbance).

Supportive Care Measures:

* G-CSF 5 mcg/kg (actual body weight) SQ daily beginning day 14. The dose will be increased to 10 mcg/kg when WBC > 1000/uL is achieved. G-CSF 10 mcg/kg should then be continued until the peripheral blood stem cell collection has been completed. All G-CSF doses should be rounded up to a convenient dose based on vial sizes of 300 and 480mcg.
* Fluoromethalone 0.1% ophthalmic solution (or equivalent medication) 2 drops qid to each eye Days 1-6.
* Voriconazole 200 mg PO Q12 hours beginning the day after completion of chemotherapy (Day +6). Equivalent anti-fungal prophylaxis with itraconazole, posaconazole or Liposomal-based amphotericin (1mg/kg) may be used.
* Patients should be hospitalized in private rooms when possible.
* Strict low bacteria diet should be used when ANC < 500 cells/uL.
* Recommended mouth care:

  a. Salt and soda swish tid
* Transfusions: Institution standards should be followed for blood product support. In lieu of standards, packed RBCes should be given to maintain the hemoglobin >8.5 gm/dl or hematocrit >25%. Platelet should be transfused to keep the platelet count >10-20 x 109/l. Blood should be filtered and irradiated (3000 cGy). CMV seronegative patients should receive CMV-seronegative blood products if available.

PERIPHERAL BLOOD STEM CELL (PBSC) COLLECTION

* Begin collections when the total white blood count exceeds 10,000/µl or when appropriate based on peripheral CD34 cell counts (institutional standard)
* Aim for a total of 1-4 collections with a standard target CD34 cell dose of > 5 x 10 x 106/kg and an optimal target CD34 cell dose of > 10 x 106/kg. The minimum CD34 cell dose is > 3 x 106/kg. Collections should continue until 10 x 106/kg CD34 (+) cell dose is achieved unless not clinically feasible.
* Stem Cell Collection: Process 18-20 L of whole blood over 3-4 hours according to institutional standards.
* PBSC Processing: The buffy coat is concentrated by centrifugation on Beckman centrifuge. Cells are suspended in Normasol media with 5% autologous plasma and 10% DMSO to a final cell concentration of 2.5 x 108/ml. Seventy ml aliquots are placed in polyolefin bags and frozen in a controlled rate freezer. Bags are labeled then stored in the liquid phase of a liquid nitrogen freezer. Institutional standard for PBSC processing should be followed.
* Four 2 ml aliquots of PBSC will be frozen in liquid nitrogen for future analysis.

TREATMENT: STEP 2 - AUTOLOGOUS STEM CELL TRANSPLANT

* Mandatory Recovery Period: The patient may begin preparative therapy for stem cell transplant following a minimum of four weeks "out-of-hospital" time since discharge from consolidation/mobilization chemotherapy.
* Dose-Adjusted Busulfan

  1. Busulfan dose should be calculated using the corrected weight which equals ideal weight + 25% of the difference between actual and ideal weight. If the actual weight is less than ideal weight use actual weight.
  2. The initial dose of busulfan (Dose cohort #1 = 1 mg/kg, Dose cohort #2 = 1.2 mg/kg, Dose cohort # 3 = 1.4) will be given as a single intravenous dose on Day -10 (in the morning, at 9:00AM). The dose will be administered by intravenous injection over 2 hours in the Outpatient Ambulatory Care/Infusion Center.

     1. The infusion tubing will be primed with busulfan diluted with saline to ensure complete administration over 2 hours as detailed in Appendix 10.
     2. The busulfan will be administered through a well functioning central venous catheter. The busulfan infusion tubing should be connected directly to the central venous catheter hub (i.e. directly to the catheter) to ensure busulfan administration over two hours.
     3. Busulfan levels will de drawn at 2, 3, 4 and 6 hours from the start of Busulfan Dose #1. For Doses #4 and #12, levels will be drawn just prior to infusion and at 2, 3, 4 and 6 hours, from a well functioning peripheral IV. (SEE Appendix 9 for busulfan sampling)
* After the busulfan is administered on Day -10, and the serial serum samples have been obtained, the patient will be discharged from the ACC infusion center.
* Busulfan dosing will resume starting on day -8 and will be given IV q6h for an additional 15 doses (total 16 doses). Patients at UCSF will receive busulfan chemotherapy on the 11 Long Adult Inpatient Unit. Dose #2 will be administered at approximately 8 pm. This dose will be adjusted based on target dose level and PK data results following dose #1. The second dose will not be given until the PK data is available from dose #1.
* PK studies will also be performed following the 4th and 12th doses. The final busulfan dose-adjustment will be made at approximately dose #10 as determined by PK data. In some cases, the dose-adjustment may be delayed due to travel time or problems at the reference lab. No dose-adjustment will be made from data obtained from samplings made following the 12th dose.
* Dose adjustments will be based on a standard formula as recommended by the reference laboratory. Adjustments will be made to achieve the target AUC level from doses 2 until 16. Dose adjustments will be calculated and confirmed by two physicians (including one of the co-PI's, if possible) at UCSF Medical Center.

Dose adjustments and busulfan laboratory values will also be reviewed regularly by Jeanine McCune Ph D., at the University of Washington, in Seattle, WA. Dr. McCune is a collaborator on this trial and manages the Busulfan pharmacokinetics laboratory in Seattle. She is a leader in the field of Busulfan metabolism, pharmacokinetics and administration.

ELIGIBILITY:
Inclusion Criteria:

Before Consolidation Chemotherapy

* Age 18-69 years
* Diagnosis of AML
* CR with ≤2 courses of induction chemotherapy.
* Out of the hospital for a minimum of 4 weeks from induction chemotherapy or 3 weeks if consolidation chemotherapy has been administered.
* Remission bone marrow bx w/i 2 wks of beginning post remission rx.
* One cycle of post-remission consolidation w/standard dose cytarabine or HDAC with <8 doses of HDAC.
* Benign CSF: Lumbar puncture with cell count, differential and protein to determine lack of extramedullary leukemia required w/i 2 weeks of post- remission therapy IF CSF status is unknown or has been positive at dx.
* No active infection
* No evidence of prior liver disease.
* Creatinine <2.0 mg/dl.
* Cardiac ejection fraction ≥40%.
* Adequate pulmonary function with DLCO ≥40% of predicted.
* No co-morbid medical condition that would jeopardize the chance of tolerating aggressive chemotherapy.
* ECOG 0-2
* Signed informed consent.

Eligibility to be Re-assessed Before Autologous SCT

* Minimum of 4 weeks out of hospital after post-remission rx.
* Continued CR documented by bone marrow morphology and cytogenetics (if previously abnormal), performed within 2 wks of admission for autologous transplantation.
* Adequate marrow recovery from post-remission therapy as demonstrated by an ANC ≥ 500/µl, platelets ≥ 50,000/µl and stable or improving hemoglobin (transfusion independent).
* Adequate peripheral stem cells collected and stored;
* No evidence of liver dysfunction as determined within 2 weeks of transplant admission. Bilirubin must be < 2.0 mg/dl and the AST and alkaline phosphatase < 3x the upper limit of normal.
* Creatinine < 2.0 mg/dl.
* No active infection or need for ongoing antibiotics.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-11; Primary Completion 2013-12-31 (Actual); Study Completion 2015-02-25 (Actual)

PRIMARY OUTCOMES:
to determine MTD amongst 3 targeted dose levels of IV busulfan given with etoposide as prep therapy in pts with AML undergoing autologous stem cell transplantation. Safety is the primary goal. | 3 yrs

SECONDARY OUTCOMES:
To achieve targeted busulfan levels following dose-adjustment of approximately (+/-) 10% in >80% of patients (i.e. target=1250 uMol*min, acceptable range 1125-1375 uMol*min, target=1400 uMol*min, acceptable range 1260-1540 ng/ml, etc) | 3 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Martin, MD, Study Chair — University of California Med. Center, SF
Locations (1):
- University of California Med. Center, San Francisco, California, United States